CLINICAL TRIAL: NCT02921516
Title: Growing Up: Intervening With HIV-Positive Adolescents in Resource-Poor Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, jessy g devieux, Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NIMH R34MH107335
Record Dates: First submitted 2016-09-24; First posted 2016-10-03 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: HIV Infection
Keywords: Adolescence; Adherence
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- N'ap Grandi (Experimental): Both Adolescent and Caregiver participate in assessment and intervention groups. Adolescent assessments will be administered at baseline, 3 months- and 6 months-post intervention. Caregiver assessments will be administered at baseline and 6 months-post intervention.
  Interventions: Behavioral: N'ap Grandi
- N'ap Grandi - A (Active Comparator): Adolescents participate in assessment and intervention groups, Caregivers participate in assessment only. Adolescent assessments will be administered at baseline, 3 months- and 6 months-post intervention. Caregiver assessments will be administered at baseline and 6 months-post intervention.
  Interventions: Behavioral: N'ap Grandi - A
- Health Promotion - A (Placebo Comparator): Adolescents participate in assessment and intervention groups, Caregivers participate in assessment only. Adolescent assessments will be administered at baseline, 3 months- and 6 months-post intervention. Caregiver assessments will be administered at baseline and 6 months-post intervention.
  Interventions: Behavioral: Health Promotion - A

INTERVENTIONS:
Behavioral: N'ap Grandi — Eight 90-minute adolescent cognitive behavioral modules and four 90-minute caregiver cognitive behavioral modules, delivered in weekend workshops over a 1 month period, with the last two modules for joint participation of adolescents and caregivers.
  Arms: N'ap Grandi
Behavioral: N'ap Grandi - A — Eight 90-minute adolescent cognitive behavioral modules delivered in weekend workshops over a 1 month period.
  Arms: N'ap Grandi - A
Behavioral: Health Promotion - A — Eight 90-minute adolescent health promotion modules delivered in weekend workshops over a 1 month period.
  Arms: Health Promotion - A

SUMMARY:
Despite overall declines in HIV incidence and mortality since ART scale-up in low and middle income countries, both have risen among youth. In addition, HIV-infected youth achieve inferior treatment outcomes compared to their adult counterparts in both high- and low-income countries, and these poorer outcomes are generally attributed to suboptimal adherence. Thus, there is a critical need for the development of adherence and risk reduction interventions for the growing cohort of these youth, and the proposed cognitive behavioral N'ap Grandi is one such intervention.

DETAILED DESCRIPTION:
As pediatric HIV infection has shifted from being a fatal disease to a chronic illness, a growing cohort of young people are moving through adolescence with all the challenges of the adult HIV-infected population but largely without comparable treatment outcomes or an evidence base to improve adherence to antiretroviral treatment (ART) and preventive behavior. Despite overall declines in HIV incidence and mortality since the ART scale-up, both have risen among youth. The goal of the proposed 3-year R34 developmental study is to respond to this need for tailored research, in particular among HIV+ older adolescents, and contribute to understanding the added value in resource-limited settings of including caregivers in an adherence and risk reduction program. Although caregiver involvement is a recognized correlate of outcomes in HIV+ youth, there are no rigorous studies of the role of caregivers in outcomes among HIV+ older adolescents.This project will integrate caregiver involvement and cognitive behavioral intervention (CBI) elements to improve ART adherence and HIV risk reduction for HIV+ older adolescents treated in resource-poor clinical settings.Our proposed study population will include caregivers and 15 to 19 year-old HIV+ youth who know their status and are receiving ART in Port-au-Prince, Haiti. Guided by the theoretical framework of the developmentally sensitive Information-Motivation-Behavioral Skills for Pediatric Adherence (IMB-PED), we will develop Growing Up (N'ap Grandi, in Haitian Creole) as a collaborative model of caregiver-adolescent engagement in the key informational, motivational, and behavioral skills antecedents of ART adherence and risk reduction. The study will utilize qualitative and quantitative methods to: identify barriers and facilitators to adherence and risk reduction (Aim 1); develop and pretest N'ap Grandi, including developmentally-appropriate manuals, training materials, procedures, and psychometric adequacy of measures (Aim 2); and assess feasibility and preliminary efficacy in a 3-arm randomized controlled trial (RCT), in which 120 youth will be assigned to three groups: the experimental caregiver-adolescent N'ap Grandi, an adolescent-only version (N'ap Grandi-A) and an adolescent-only health promotion group (HP-A), examining ART adherence and virologic response, HIV risk behaviors, positive communication and monitoring, stress and mood, and costs from the health center perspective (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

1. youth aged 15-19 years receiving 1st-line ART for at least 3 months;
2. exhibiting risk factors of detectable Viral Load and/or unprotected vaginal/anal intercourse in the previous 6 months;
3. fluent in spoken Haitian Creole which is required to complete assessments and to participate in the intervention groups;
4. willing to a) assent to study participation if under 18, and b) having a parent or caregiver aged >18 years provide informed consent and participate in the caregiver workshops.

Exclusion Criteria:

1. cognitively impaired, as determined by the Test of Nonverbal Intelligence (TONI), since such impairment may compromise the ability to comprehend and participate in the assessment and intervention;
2. exhibits bipolar disorder, psychosis, or current need for inpatient psychiatric hospitalization.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 278 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
ART Adherence and response | 6 months
  Data from self report questionnaire (percent medications taken), medication possession ratio (percent completed), and virologic suppression (percent improvement) will be aggregated into a composite measure of adherence.

SECONDARY OUTCOMES:
HIV sexual transmission risk reduction | 6 months
  Increase in self-reported safer sex behavior via questionnaire
Caregiver supportive communication | 6 months
  Increase in self-reported positive caregiver-adolescent communication and monitoring via questionnaire
Psychosocial health | 6 months
  Improvement in self-reported stress and mood via questionnaire
Cost of intervention from the health center perspective | 6 months
  Provide data on the economic feasibility of broader scale up of these interventions

CONTACTS AND LOCATIONS:
Overall Officials: Jessy G. Dévieux, Ph.D., Principal Investigator — Florida International University
Locations (1):
- GHESKIO Centers, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: No